CLINICAL TRIAL: NCT04456699
Title: A Phase 3 Randomized, Open-label Study to Evaluate the Efficacy and Safety of Olaparib Alone or in Combination With Bevacizumab Compared to Bevacizumab With a Fluoropyrimidine in Participants With Unresectable or Metastatic Colorectal Cancer Who Have Not Progressed Following First-line Induction (LYNK-003)
Brief Title: Efficacy and Safety of Olaparib (MK-7339) With or Without Bevacizumab Compared to Bevacizumab With a Fluoropyrimidine in Unresectable or Metastatic Colorectal Cancer (CRC) (MK-7339-003/LYNK-003)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7339-003; MK-7339-003 (Other: MSD); LYNK-003 (Other: MSD); jRCT2031200146 (Registry Identifier: jRCT); 2019-000698-22 (EudraCT Number)
Record Dates: First submitted 2020-07-01; First posted 2020-07-02 (Actual); Results first posted 2024-04-02 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Metastatic Colorectal Cancer
Keywords: colorectal cancer; CRC; Olaparib; Bevacizumab; FOLFOX; 5-FU; fluorouracil; folinic acid; oxaliplatin; CAPOX; capecitabine
MeSH Terms: conditions — Colorectal Neoplasms | interventions — olaparib; Fluorouracil; Bevacizumab; Capecitabine; Leucovorin; Levoleucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Olaparib + bevacizumab (Experimental): Participants will receive olaparib (300 mg twice daily [BID] oral) + Bevacizumab (5 mg/kg intravenous [IV] once every 2 weeks [Q2W]) until progressive disease or end of study.
  Interventions: Drug: Olaparib; Drug: Bevacizumab
- Olaparib (Experimental): Participants will receive olaparib (300 mg BID) oral, until progressive disease or end of study.
  Interventions: Drug: Olaparib
- Bevacizumab + chemotherapy (Active Comparator): Participants will receive investigator's choice of either bevacizumab (7.5 mg/kg IV once every three weeks (Q3W)) + capecitabine (1000 mg/m^2 BID for 14 days, then 7 days off, Q3W) or bevacizumab (5 mg/kg IV Q2W) + 5-FU (2400 mg/m2 IV over 46 to 48 hours Q2W; bolus 5-FU (400 mg/m2) can be added prior to infusional 5-FU, per local standards and at the investigator's discretion). Leucovorin or levoleucovorin 400 mg/m^2 (leucovorin) or 200 mg/m^2 (levoleucovorin) Q2W IV infusion may be added per investigator's discretion. Treatment will continue until progressive disease or end of study.
  Interventions: Drug: 5-FU; Drug: Bevacizumab; Drug: Capecitabine; Drug: Leucovorin/ levoleucovorin

INTERVENTIONS:
Drug: Olaparib — 300 mg BID, oral until progressive disease or end of study
  Other Names: LYNPARZA^TM
  Arms: Olaparib; Olaparib + bevacizumab
Drug: 5-FU — 2400 mg/m^2 over 46 to 48 hours Q2W IV infusion until disease progression or end of study; bolus 5-FU (400mg/m2) can be added prior to infusional 5-FU, per local standards and at the investigator's discretion
  Other Names: Fluorouracil; Adrucil; Efudex
  Arms: Bevacizumab + chemotherapy
Drug: Bevacizumab — 5 mg/kg or 7.5 mg/kg Q2W or Q3W IV infusion until progressive disease or end of study
  Other Names: MVASI^TM; Avastin
  Arms: Bevacizumab + chemotherapy; Olaparib + bevacizumab
Drug: Capecitabine — 1000 mg/m^2 oral capsule BID for 14 days, then 7 days off, Q3W) until progressive disease or end of study
  Other Names: XELODA^®
  Arms: Bevacizumab + chemotherapy
Drug: Leucovorin/ levoleucovorin — 400 mg/m^2 (leucovorin) or 200 mg/m^2 (levoleucovorin) may be added to Bevacizumab + 5-FU per investigator's discretion Q2W IV infusion until progressive disease or end of study
  Other Names: Folinic Acid; Fusilev^®; Khapzory^TM
  Arms: Bevacizumab + chemotherapy

SUMMARY:
This is an efficacy and safety study of olaparib alone or in combination with bevacizumab being compared to bevacizumab with a fluoropyrimidine in participants with unresectable or metastatic colorectal cancer who have not progressed following first-line induction. The primary hypotheses are: Olaparib + Bevacizumab is superior to a fluoropyrimidine + Bevacizumab with respect to progression-free survival (PFS) using Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST 1.1) as assessed by blinded independent central review (BICR); Olaparib is superior to a fluoropyrimidine + Bevacizumab with respect to PFS using RECIST 1.1 as assessed by BICR. As of amendment 5 study enrollment is being discontinued and study participants randomized to one of the two experimental arms (olaparib plus bevacizumab or olaparib monotherapy) must discontinue study intervention. Participants who are still on study treatment will no longer have tumor response assessments by BICR.

ELIGIBILITY:
Inclusion Criteria:

1. Has a histologically-confirmed metastatic or unresectable (Stage IV as defined by American Joint Committee on Cancer (AJCC eighth edition) colorectal adenocarcinoma (National Comprehensive Cancer Network [NCCN] 2018).
2. Has not progressed (ie, achieved a stable disease [SD], partial response [PR], or complete response [CR]) after a first-line induction course of at least 6 cycles of folinic acid/fluorouracil/oxaliplatin (FOLFOX) + bevacizumab or 4 cycles of capecitabine and oxaliplatin (CAPOX) + bevacizumab as first-line therapy.

   * Participants must not have received an investigational agent during their induction course.
   * Determination of best overall response (SD/PR/CR) will be made by the investigator.
   * Non-Progressive Disease (PD) will be verified by BICR prior to randomization based on the images submitted to imaging contract research organization (iCRO) as described in inclusion criterion 4.
   * "First-line therapy" is defined as the first systemic chemotherapy regimen given for the diagnosis of unresectable or metastatic colorectal cancer (CRC). Participants may have received prior adjuvant/neoadjuvant chemotherapy for CRC, as long as it was completed at least 6 months prior to initiation of first-line CAPOX + bevacizumab or FOLFOX + bevacizumab induction treatment.
3. Has experienced unacceptable toxicity to oxaliplatin that, in the opinion of the treating physician, requires/required the discontinuation of oxaliplatin. Note: As an example, unacceptable toxicity may include (but is not limited to) severe or prolonged neurotoxicity.

   • Participants must be randomized within a minimum of 2 weeks and a maximum of 6 weeks after their last dose of CAPOX + bevacizumab or FOLFOX + bevacizumab (last dose is the day of the last infusion that contained oxaliplatin).
4. Has provided to the iCRO 1 set of baseline radiographic images taken before or during the CAPOX + bevacizumab or FOLFOX + bevacizumab induction period and at least 42 days prior to the imaging performed during Screening. Tumor imaging at Screening must be performed within 28 days prior to the date of randomization.
5. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 within 10 days prior to randomization.

Exclusion Criteria:

1. Has known hypersensitivity to the components and/or excipients in bevacizumab, 5-FU, capecitabine, or olaparib.
2. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable (ie, without evidence of progression for at least 28 days by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid intervention for at least 14 days prior to first dose of study intervention.
3. Has an active infection requiring systemic therapy.
4. Has a known history of human immunodeficiency virus (HIV) infection. No HIV testing is required unless mandated by local health authority.
5. Has a known history of or is positive for hepatitis B surface antigen (HBsAg reactive) or hepatitis C ribonucleic acid (HCV RNA [qualitative]) is detected). Note: No testing for hepatitis B and hepatitis C is required unless mandated by local health authority.
6. Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study.
7. Has myelodysplastic syndrome/acute myeloid leukemia (MDS/AML) or with features suggestive of MDS/AML.
8. Has hemoptysis or hematemesis within 28 days prior to randomization.
9. Has evidence of bleeding diathesis or significant coagulopathy (in the absence of anticoagulation).
10. Has clinically significant bleeding within 28 days prior to randomization.
11. Is considered a poor medical risk due to a serious, uncontrolled medical disorder, nonmalignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on high-resolution computed tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent.
12. Has 1 or more conditions that, in the opinion of the treating physician, make the participant ineligible for treatment with bevacizumab. These conditions may include:

    * Uncontrolled hypertension (systolic blood pressure [SBP] >150 mm Hg or diastolic blood pressure [DBP] >100 mm Hg) or a history of hypertensive crisis or hypertensive encephalopathy
    * Arterial thromboembolic events (eg, myocardial infarction, cerebral infarction)
    * History of nephrotic syndrome or moderate proteinuria
    * History of gastrointestinal perforation
    * History of non-gastrointestinal fistula formation
    * History of possible reversible encephalopathy syndrome (RPLS)
13. Has received prior systemic anticancer therapy (other than CAPOX + bevacizumab or FOLFOX + bevacizumab induction) including investigational agents within 28 days prior to randomization. Note: Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with persistent alopecia or Grade ≤3 neuropathy are eligible.
14. Has received prior therapy with olaparib or with any other polyadenosine 5'-diphosphoribose polymerase (PARP) inhibitor.
15. Is currently receiving either strong (eg, itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate (eg, ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil) inhibitors of cytochrome P450 3A4 (CYP3A4) that cannot be discontinued for the duration of the study. The required washout period prior to randomization is 2 weeks.
16. Is currently receiving either strong (phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate (eg. bosentan, efavirenz, modafinil) inducers of CYP3A4 that cannot be discontinued for the duration of the study. The required washout period prior to randomization is 5 weeks for phenobarbital and 3 weeks for other agents.
17. Has undergone major surgery within 2 weeks of randomization or has not recovered adequately from toxicities and/or complications from any major surgery prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 335 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (129):
- United States (23):
  - Providence Saint Joseph Medical Center, Disney Family Cancer ( Site 1392), Burbank, California
  - St Joseph Heritage Healthcare-Oncology ( Site 1383), Fullerton, California
  - UC Health Memorial Hospital ( Site 1401), Colorado Springs, Colorado
  - Poudre Valley Health System ( Site 1402), Fort Collins, Colorado
  - University Cancer & Blood Center, LLC ( Site 1381), Athens, Georgia
  - University of Chicago ( Site 1357), Chicago, Illinois
  - Illinois Cancer Care, PC ( Site 1352), Peoria, Illinois
  - James Graham Brown Cancer Center ( Site 1393), Louisville, Kentucky
  - University Medical Center New Orleans ( Site 1365), New Orleans, Louisiana
  - New England Cancer Specialists ( Site 1422), Scarborough, Maine
  - Cancer & Hematology Centers of Western Michigan ( Site 1358), Grand Rapids, Michigan
  - Hattiesburg Clinic Hematology/Oncology ( Site 1418), Hattiesburg, Mississippi
  - Washington University in St. Louis ( Site 1384), St Louis, Missouri
  - St. Vincent Frontier Cancer Center-Research ( Site 1414), Billings, Montana
  - CHI Health St. Francis ( Site 1406), Grand Island, Nebraska
  - Cancer Partners of Nebraska ( Site 1353), Lincoln, Nebraska
  - Providence Portland Medical Center ( Site 1400), Portland, Oregon
  - Oregon Health & Science University ( Site 1411), Portland, Oregon
  - Allegheny Singer Research Institute ( Site 1364), Pittsburgh, Pennsylvania
  - West Cancer Center - East Campus ( Site 1396), Germantown, Tennessee
  - Vanderbilt University Medical Center ( Site 1362), Nashville, Tennessee
  - Baylor Scott & White Medical Center - Temple ( Site 1397), Temple, Texas
  - Blue Ridge Cancer Care ( Site 1374), Roanoke, Virginia
- Australia (6):
  - St George Hospital ( Site 0052), Kogarah, New South Wales
  - Liverpool Hospital ( Site 0055), Liverpool, New South Wales
  - Royal Brisbane and Women s Hospital ( Site 0054), Herston, Queensland
  - Queen Elizabeth Hospital ( Site 0053), Woodville South, South Australia
  - Monash Health ( Site 0050), Clayton, Victoria
  - Peninsula Health Frankston Hospital ( Site 0056), Frankston, Victoria
- Belgium (8):
  - Imelda vzw ( Site 0110), Bonheiden, Antwerpen
  - AZ Klina ( Site 0106), Brasschaat, Antwerpen
  - UZ Antwerpen ( Site 0108), Edegem, Antwerpen
  - UCL Saint Luc ( Site 0100), Brussels, Bruxelles-Capitale, Region de
  - OLV Ziekenhuis ( Site 0109), Aalst, Oost-Vlaanderen
  - UZ Gent ( Site 0101), Ghent, Oost-Vlaanderen
  - UZ Gasthuisberg ( Site 0102), Leuven, Vlaams-Brabant
  - AZ Groeninge ( Site 0105), Kortrijk, West-Vlaanderen
- Canada (6):
  - Dr. Everett Chalmers Regional Hospital ( Site 0204), Fredericton, New Brunswick
  - Moncton Hospital - Horizon Health Network ( Site 0201), Moncton, New Brunswick
  - Princess Margaret Cancer Centre ( Site 0209), Toronto, Ontario
  - Hopital Cite de la Sante de Laval ( Site 0203), Laval, Quebec
  - McGill University Health Centre ( Site 0207), Montreal, Quebec
  - CIUSSS de l Estrie - CHUS - Centre Hosp. Univ. Sherbrooke ( Site 0202), Sherbrooke, Quebec
- Chile (3):
  - Sociedad Oncovida S.A. ( Site 0250), Santiago, Region M. de Santiago
  - Clínica San Carlos de Apoquindo Red Salud UC Christus ( Site 0252), Santiago, Region M. de Santiago
  - Centro Investigación del Cáncer James Lind ( Site 0251), Temuco, Región de la Araucanía
- Colombia (7):
  - Administradora Country SA - Clinica del Country ( Site 0350), Bogotá, Bogota D.C.
  - Instituto Nacional de Cancerologia E.S.E ( Site 0362), Bogotá, Bogota D.C.
  - Sociedad de Oncología Y Hematología del Cesar S.A.S. ( Site 0353), Valledupar, Cesar Department
  - Oncomedica S.A. ( Site 0352), Montería, Departamento de Córdoba
  - Oncologos del Occidente ( Site 0364), Pereira, Risaralda Department
  - Fundacion Cardiovascular de Colombia ( Site 0360), Bucaramanga, Santander Department
  - Hemato Oncologos S.A. ( Site 0355), Cali, Valle del Cauca Department
- France (7):
  - Centre Leon Berard ( Site 0459), Lyon, Auvergne-Rhône-Alpes
  - C.H.U. de Strasbourg Hopital de Hautepierre ( Site 0464), Strasbourg, Bas-Rhin
  - Institut de Cancerologie de l Ouest Centre Rene Gauducheau ( Site 0455), Saint-Herblain, Brittany Region
  - CHU Jean Minjoz ( Site 0450), Besançon, Doubs
  - CHU Bordeaux Haut-Leveque ( Site 0457), Pessac, Gironde
  - CHU Saint Eloi ( Site 0467), Montpellier, Herault
  - Hopital Europeen Georges Pompidou ( Site 0452), Paris
- Germany (4):
  - Universitaetsklinikum Ulm ( Site 0500), Ulm, Baden-Wurttemberg
  - St. Josef und St. Elisabeth Hospital gGmbH-Hematology, oncology and palliative medicine ( Site 0503), Bochum, North Rhine-Westphalia
  - Charité Universitaetsmedizin Berlin - Campus Mitte ( Site 0504), Berlin
  - Facharztzentrum Eppendorf ( Site 0501), Hamburg
- Hungary (6):
  - Bekes Megyei Kozponti Korhaz - Pandy Kalman Tagkorhaza ( Site 1432), Gyula, Bekes County
  - Borsod-Abaúj-Zemplén Megyei Központi Kórház és Egyetemi Okta-Klinikai Onkológiai és Sugárterápiás Ce, Miskolc, Borsod-Abauj Zemplen county
  - Debreceni Egyetem Klinikai Kozpont ( Site 1426), Debrecen, Hajdú-Bihar
  - Jasz Nagykun Szolnok Megyei Hetenyi Geza Korhaz Rendelointezet ( Site 1427), Szolnok, Jász-Nagykun-Szolnok
  - Zala Megyei Szent Rafael Korhaz ( Site 1429), Zalaegerszeg, Zala County
  - Orszagos Onkologiai Intezet ( Site 1431), Budapest
- Japan (10):
  - Aichi Cancer Center Hospital ( Site 0658), Nagoya, Aichi-ken
  - National Cancer Center Hospital East ( Site 0650), Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center ( Site 0652), Matsuyama, Ehime
  - St. Marianna University School of Medicine Hospital ( Site 0657), Kawasaki, Kanagawa
  - Saitama Cancer Center ( Site 0653), Kitaadachi-gun, Saitama
  - Shizuoka Cancer Center Hospital and Research Institute ( Site 0655), Sunto-gun, Shizuoka
  - Chiba Cancer Center ( Site 0656), Chiba
  - National Hospital Organization Kyushu Cancer Center ( Site 0654), Fukuoka
  - National Cancer Center Hospital ( Site 0651), Tokyo
  - The Cancer Institute Hospital of JFCR ( Site 0659), Tokyo
- Latvia (3):
  - Daugavpils Regional Hospital ( Site 1502), Daugavpils
  - P. Stradina Clinical University Hospital ( Site 1500), Riga
  - Riga East Clinical University Hospital ( Site 1501), Riga
- Lithuania (3):
  - LSMUL Kauno Klinikos ( Site 1528), Kaunas
  - Nacionalinis Vezio Institutas ( Site 1527), Vilnius
  - Vilniaus Universiteto Ligonine Santaros Klinikos ( Site 1526), Vilnius
- Russia (9):
  - Arkhangelsk Clinical Oncological Dispensary ( Site 1113), Arkhangelsk, Arkhangelskaya oblast
  - GBUZ Republican Clinical Oncological Dispensary-Antitumor drug therapy department ( Site 1130), Ufa, Baskortostan, Respublika
  - Krasnoyarsk Regional Clinical Oncological Dispensary ( Site 1121), Krasnoyarsk, Krasnoyarsk Krai
  - National Medical and Surgical Center n.a. N.I.Pirogov ( Site 1126), Moscow, Moscow
  - N.N. Blokhin NMRCO ( Site 1106), Moscow, Moscow
  - First Moscow State Medical University n.a. I.M.Sechenov ( Site 1127), Moscow, Moscow
  - MROI n.a. P.A. Herzen - branch of FSBI NMICR of MoH of Russia ( Site 1128), Moscow, Moscow
  - MEDSI Clinical Hospital on Pyatnitsky Highway-Departmentof Antitumor Drug therapy ( Site 1129), Krasnogorsk, Moscow Oblast
  - City Clinical Oncology Center ( Site 1114), Saint Petersburg, Sankt-Peterburg
- South Africa (3):
  - Sandton Oncology Medical Group PTY LTD ( Site 0900), Sandton, Gauteng
  - The Oncology Centre ( Site 0903), Durban, Limpopo
  - Cancercare Rondebosch Oncology ( Site 0904), Rondebosch, Western Cape
- South Korea (7):
  - Asan Medical Center ( Site 0952), Songpagu, Seoul
  - Kyungpook National University Chilgok Hospital ( Site 0956), Daegu, Taegu-Kwangyokshi
  - Korea University Anam Hospital ( Site 0955), Seoul
  - Seoul National University Hospital ( Site 0950), Seoul
  - Severance Hospital Yonsei University Health System ( Site 0951), Seoul
  - Samsung Medical Center ( Site 0954), Seoul
  - The Catholic University of Korea St. Mary s Hospital ( Site 0953), Seoul
- Spain (5):
  - Hospital General Universitario de Elche ( Site 1155), Elche, Alicante
  - Hospital Universitario Central de Asturias ( Site 1153), Oviedo, Principality of Asturias
  - Hospital Vall D Hebron ( Site 1151), Barcelona
  - Hospital Universitario Gregorio Maranon ( Site 1152), Madrid
  - Hospital 12 de Octubre de Madrid ( Site 1150), Madrid
- Turkey (Türkiye) (11):
  - Inonu Universitesi Medical Fakultesi ( Site 1207), Malatya, Adana
  - Baskent University Adana Training Hospital ( Site 1205), Adana
  - Hacettepe University Faculty of Medicine ( Site 1200), Ankara
  - Gazi Universitesi Tip Fakultesi ( Site 1215), Ankara
  - Trakya Universitesi Tip Fakultesi ( Site 1210), Edirne
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi ( Site 1202), Istanbul
  - Prof. Dr. Cemil Tascioglu Sehir Hastanesi ( Site 1216), Istanbul
  - Göztepe Prof. Dr. Süleyman Yalçın Şehir Hastanesi-oncology ( Site 1214), Istanbul
  - Kartal Dr. Lutfi Kirdar Egitim ve Arast Hast ( Site 1211), Istanbul
  - Ege Universitesi Tip Fakultesi Tulay Aktas Onkoloji Hastanesi ( Site 1204), Izmir
  - Necmettin Erbakan Universitesi Meram Tip Fakultesi ( Site 1203), Konya
- Ukraine (8):
  - Medical center Medikal Plaza of Ecodnipro LLC ( Site 1317), Dnipro, Dnipropetrovsk Oblast
  - Communal non profit enterprise Regional Clinical Oncology Center ( Site 1304), Kharkiv, Kharkivs’ka Oblast’
  - Medical Center of Yuriy Spizhenko LLC.-Clinical Trial ( Site 1319), Kapitanivka Village, Kyivska Oblast
  - Medical Center Asklepion LLC ( Site 1309), Khodosovka, Kyivska Oblast
  - Medical Center Verum ( Site 1318), Kyiv, Kyivska Oblast
  - Shalimov s NI of Surgery and Transplantation ( Site 1321), Kyiv, Kyivska Oblast
  - Medical center of the Limited Liability Company Yulis ( Site 1314), Zaporizhzhia, Zaporizhzhia Oblast
  - Dobrobut Medical Center ( Site 1320), Kyiv

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Takashima A, Garcia-Alfonso P, Manneh R, Besen AA, Hong YS, Cuyle PJ, Yanez P, Burge M, Yoshino T, Kim TW, Cui K, Li C, Jain R, Adelberg D, Taieb J. Olaparib with or without bevacizumab versus bevacizumab plus a fluoropyrimidine as maintenance therapy in advanced colorectal cancer: The randomized phase 3 LYNK-003 study. Eur J Cancer. 2024 Jul;205:114036. doi: 10.1016/j.ejca.2024.114036. Epub 2024 Mar 21. PMID 38749110
- [Derived] Kim TW, Taieb J, Gurary EB, Lerman N, Cui K, Yoshino T. Olaparib with or without bevacizumab or bevacizumab and 5-fluorouracil in advanced colorectal cancer: Phase III LYNK-003. Future Oncol. 2021 Dec;17(36):5013-5022. doi: 10.2217/fon-2021-0899. Epub 2021 Nov 15. PMID 34779646
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26089&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible participants were randomized 1:1:1 to receive either Olaparib + Bevacizumab, Olaparib, or Bevacizumab + chemotherapy.
Groups:
- Olaparib + Bevacizumab: Participants received olaparib (300 mg twice daily [BID] oral) + Bevacizumab (5 mg/kg intravenous [IV] once every 2 weeks [Q2W]) until progressive disease or end of study.
- Olaparib: Participants received olaparib (300 mg BID) oral, until progressive disease or end of study.
- Bevacizumab + Chemotherapy: Participants received investigator's choice of either bevacizumab (7.5 mg/kg IV once every three weeks (Q3W)) + capecitabine (1000 mg/m^2 BID for 14 days, then 7 days off, Q3W) or bevacizumab (5 mg/kg IV Q2W) + 5-FU (2400 mg/m2 IV over 46 to 48 hours Q2W; bolus 5-FU (400 mg/m2) was added prior to infusional 5-FU, per local standards and at the investigator's discretion). Leucovorin or levoleucovorin 400 mg/m^2 (leucovorin) or 200 mg/m^2 (levoleucovorin) Q2W IV infusion was added per investigator's discretion. Treatment continued until progressive disease or end of study.
Period: Overall Study
Arm/Group | Olaparib + Bevacizumab | Olaparib | Bevacizumab + Chemotherapy
Started | 111 | 115 | 109
Treated | 111 | 113 | 108
Completed | 0 | 0 | 0
Not Completed | 111 | 115 | 109
Not completed — Death | 48 | 50 | 52
Not completed — Physician Decision | 0 | 0 | 2
Not completed — Sponsor Decision | 55 | 61 | 50
Not completed — Withdrawal by Subject | 8 | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olaparib + Bevacizumab | Olaparib | Bevacizumab + Chemotherapy | Total
Number analyzed (Participants) | 111 | 115 | 109 | 335
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.5 (12.8) | 61.1 (10.7) | 63.2 (11.3) | 61.3 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 49 | 44 | 143
  Male | 61 | 66 | 65 | 192
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 16 | 10 | 44
  Not Hispanic or Latino | 88 | 93 | 94 | 275
  Unknown or Not Reported | 5 | 6 | 5 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 10 | 5 | 4 | 19
  Asian | 25 | 40 | 30 | 95
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 71 | 64 | 66 | 201
  More than one race | 2 | 3 | 4 | 9
  Unknown or Not Reported | 3 | 3 | 4 | 10
Response to Prior Induction [Count of Participants; unit: Participants] — Participants last scan prior to folinic acid/fluorouracil/oxaliplatin (FOLFOX) + bevacizumab or capecitabine and oxaliplatin (CAPOX) + bevacizumab treatment was assessed by blinded independent central review (BICR) per (Response Evaluation Criteria in Solid Tumors RECIST) 1.1 criteria to evaluate presence of stable disease (SD; Neither sufficient shrinkage to qualify for partial response [PR] nor sufficient increase to qualify for progressive disease), complete response (CR; Disappearance of all target lesions) or PR (At least a 30% decrease in sum of diameters of target lesions).
  Participants
    CR/PR | 49 | 48 | 47 | 144
    SD | 62 | 67 | 62 | 191
Number of Induction Cycles [Count of Participants; unit: Participants] — Number of induction cycles received was assessed at the baseline and categorized as: 1) 6-8 cycles for FOLFOX + bevacizumab or 4-6 cycles for CAPOX + bevacizumab and 2) >8 cycles for FOLFOX + bevacizumab or >6 cycles for CAPOX + bevacizumab.
  Participants
    6-8 cycles for FOLFOX + bevacizumab or 4-6 cycles for CAPOX + bevacizumab | 53 | 57 | 53 | 163
    >8 cycles for FOLFOX + bevacizumab or >6 cycles for CAPOX + bevacizumab | 58 | 58 | 56 | 172
Mutation Status [Count of Participants; unit: Participants] — Participants were assessed for BRAF and/or Ras mutations versus wild type for both (BRAFwt + RASwt) at baseline.
  Participants
    BRAF and RAS all wild type | 32 | 33 | 29 | 94
    BRAF or RAS Mutation | 79 | 82 | 80 | 241

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version (RECIST) 1.1 as Assessed by Blinded Independent Central Review (BICR)
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions was also considered PD. PFS using RECIST 1.1 as assessed by BICR is presented.
Time Frame: Up to approximately 30 months
Population: The analysis population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib + Bevacizumab | Olaparib | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 111 | 115 | 109
Months | 3.7 [3.4 to 5.3] | 3.6 [2.0 to 3.7] | 5.5 [3.8 to 5.6]
Statistical Analysis 1: Comparison: Olaparib + Bevacizumab vs Bevacizumab + Chemotherapy; Test type: Superiority; p = 0.9774, Log Rank; One-sided p-value based on log-rank test stratified by prior FOLFOX/CAPOX + Bev induction response, number of induction cycles and mutation status; Hazard Ratio (HR) = 1.41, 95% CI 2-sided [1.00 to 1.97] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by prior FOLFOX/CAPOX + Bev induction response, number of induction cycles and mutation status
Statistical Analysis 2: Comparison: Olaparib vs Bevacizumab + Chemotherapy; Test type: Superiority; p = 0.9993, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.75, 95% CI 2-sided [1.23 to 2.49] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause. The OS is presented.
Time Frame: Up to approximately 30 months
Population: The analysis population consists of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib + Bevacizumab | Olaparib | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 111 | 115 | 109
Months | 21.2 [15.1 to NA] — NA=OS upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | 21.6 [17.2 to NA] — NA=OS upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | 19.9 [13.8 to 22.5]
Statistical Analysis 1: Comparison: Olaparib + Bevacizumab vs Bevacizumab + Chemotherapy; Test type: Superiority; p = 0.1527, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.54 to 1.21] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Olaparib vs Bevacizumab + Chemotherapy; Test type: Superiority; p = 0.2491, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.59 to 1.30] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Objective Response Rate (ORR) Per RECIST 1.1 as Assessed by BICR
Description: ORR was defined as the percentage of participants who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ.
Time Frame: Up to approximately 30 months
Population: The analysis population consisted of all randomized participants who had a measurable disease.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Olaparib + Bevacizumab | Olaparib | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 104 | 107 | 105
Percentage of Participants | 4.8 [1.6 to 10.9] | 1.9 [0.2 to 6.6] | 4.8 [1.6 to 10.8]
Statistical Analysis 1: Comparison: Olaparib + Bevacizumab vs Bevacizumab + Chemotherapy; Test type: Superiority; p = 0.5272, Miettinen and Nurminen; Based on stratified Miettinen & Nurminen method. One-sided p-value for testing H0: difference in % = 0 versus H1: difference in % > 0; Difference in Percentage = -0.2, 95% CI 2-sided [-7.0 to 6.5] — Based on Miettinen & Nurminen method stratified by prior FOLFOX/CAPOX + Bev induction response, cycles and mutation status
Statistical Analysis 2: Comparison: Olaparib vs Bevacizumab + Chemotherapy; Test type: Superiority; p = 0.9020, Miettinen & Nurminen; [statistical method as in outcome 3, analysis 1]; Difference in Percentage = -3.2, 95% CI 2-sided [-9.7 to 2.3] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Number of Participants With One or More Adverse Events (AE)
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experienced at least one AE was reported for each arm.
Time Frame: Up to approximately 30 months
Population: All randomized participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib + Bevacizumab | Olaparib | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 111 | 113 | 108
Participants | 101 | 91 | 96

5. Secondary Outcome: Number of Participants Discontinuing Study Intervention Due to an AE
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinued study intervention due to an AE was reported for each arm.
Time Frame: Up to approximately 30 months
Population: All randomized participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib + Bevacizumab | Olaparib | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 111 | 113 | 108
Participants | 6 | 4 | 7

6. Secondary Outcome: Duration of Response (DOR) Per RECIST 1.1 as Assessed by BICR
Description: For participants who demonstrate a confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. DOR is defined as the time from first documented evidence of a CR or PR until progressive disease (PD) or death. DOR for participants who had not progressed or died at the time of analysis will be censored at the date of their last tumor assessment. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions as well as an absolute increase of at least a 5 mm in the sum of diameters. The appearance of one or more new lesions is also considered PD. DOR assessments will be based on BICR with confirmation. The DOR as assessed using RECIST 1.1 for all participants who experience a confirmed CR or PR will be presented.
Time Frame: Up to approximately 30 months
Population: All randomized participants who received at least one dose of treatment and had either a CR or a PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib + Bevacizumab | Olaparib | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 5 | 2 | 5
Months | NA [3.6 to NA] — NA = Median and upper limit of 95% CI for DOR was not reached due to insufficient number of participants with a response. | NA [NA to NA] — NA = Median, lower limit, and upper limit of 95% CI for DOR was not reached due to insufficient number of participants with a response. | NA [NA to NA] — NA = Median, lower limit, and upper limit of 95% CI for DOR was not reached due to insufficient number of participants with a response.

ADVERSE EVENTS:
Time Frame: Up to approximately 38 months
Description: Serious and Other adverse events (AEs) includes all participants who received ≥1 dose of study treatment. All-Cause Mortality includes all randomized participants. Per protocol, disease progression of cancer under study was not considered an AE unless considered related to study treatment. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" & "Disease progression" not related to study treatment are excluded as AEs.
Arm/Group | Olaparib + Bevacizumab | Olaparib | Bevacizumab + Chemotherapy
All-Cause Mortality (participants affected / at risk) | 49/111 | 51/115 | 52/109
Serious Adverse Events (participants affected / at risk) | 16/111 | 13/113 | 14/108
Other Adverse Events (participants affected / at risk) | 94/111 | 74/113 | 86/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaparib + Bevacizumab (N=111) | Olaparib (N=113) | Bevacizumab + Chemotherapy (N=108)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Duodenal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Rectal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Large intestine infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Parotitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Skin candida (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (2)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Human rhinovirus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaparib + Bevacizumab (N=111) | Olaparib (N=113) | Bevacizumab + Chemotherapy (N=108)
Anaemia (Blood and lymphatic system disorders) | 32 (35) | 21 (25) | 8 (9)
Neutropenia (Blood and lymphatic system disorders) | 9 (14) | 5 (6) | 1 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (8) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 19 (22) | 8 (8) | 13 (14)
Abdominal pain upper (Gastrointestinal disorders) | 8 (9) | 4 (5) | 2 (2)
Constipation (Gastrointestinal disorders) | 16 (18) | 11 (11) | 14 (15)
Diarrhoea (Gastrointestinal disorders) | 11 (16) | 9 (9) | 15 (15)
Nausea (Gastrointestinal disorders) | 31 (38) | 23 (26) | 24 (35)
Stomatitis (Gastrointestinal disorders) | 8 (9) | 4 (4) | 11 (13)
Vomiting (Gastrointestinal disorders) | 13 (17) | 7 (13) | 11 (14)
Asthenia (General disorders) | 16 (22) | 8 (8) | 11 (14)
Fatigue (General disorders) | 14 (15) | 15 (15) | 10 (11)
Pyrexia (General disorders) | 10 (10) | 5 (5) | 7 (9)
Urinary tract infection (Infections and infestations) | 5 (6) | 4 (4) | 6 (9)
Aspartate aminotransferase increased (Investigations) | 5 (6) | 6 (7) | 6 (8)
Blood creatinine increased (Investigations) | 4 (4) | 2 (2) | 6 (9)
Neutrophil count decreased (Investigations) | 9 (20) | 7 (8) | 3 (5)
Platelet count decreased (Investigations) | 2 (3) | 6 (7) | 7 (8)
Weight decreased (Investigations) | 7 (7) | 2 (2) | 6 (6)
Decreased appetite (Metabolism and nutrition disorders) | 15 (15) | 18 (20) | 12 (13)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 10 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (13) | 7 (8) | 8 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 3 (3) | 8 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1) | 5 (7)
Dysgeusia (Nervous system disorders) | 10 (12) | 3 (4) | 3 (4)
Headache (Nervous system disorders) | 7 (7) | 1 (1) | 3 (3)
Neuropathy peripheral (Nervous system disorders) | 3 (5) | 7 (7) | 4 (4)
Proteinuria (Renal and urinary disorders) | 1 (1) | 3 (3) | 10 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 0 (0) | 4 (6)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 8 (8)
Hypertension (Vascular disorders) | 11 (12) | 0 (0) | 10 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-08): https://cdn.clinicaltrials.gov/large-docs/99/NCT04456699/Prot_SAP_001.pdf